CLINICAL TRIAL: NCT02745769
Title: An Open-Label, Phase 1a/1b Study of Ramucirumab in Combination With Other Targeted Agents in Advanced Cancers
Brief Title: A Study in Advanced Cancers Using Ramucirumab (LY3009806) and Other Targeted Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16165; I4T-MC-JVDK (Other: Eli Lilly and Company); 2015-004381-28 (EudraCT Number)
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03-01

CONDITIONS: Advanced Cancer; Colorectal Cancer; Mantle Cell Lymphoma
MeSH Terms: conditions — Colorectal Neoplasms; Lymphoma, Mantle-Cell | interventions — Ramucirumab; merestinib; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramucirumab + Merestinib (Experimental): Ramucirumab intravenously (IV) on day 1 and day 15 in combination with merestinib orally once a day over a 28 day cycle. Participants receiving benefit may continue until disease progression.
  Interventions: Drug: Ramucirumab; Drug: Merestinib
- Ramucirumab + Abemaciclib (Experimental): Ramucirumab IV on day 1 and day 15 in combination with abemaciclib orally twice a day over a 28 day cycle. Participants receiving benefit may continue until disease progression.
  On June 21st 2017 the Ramucirumab + Abemaciclib arm was cancelled with no participants enrolled.
  Interventions: Drug: Ramucirumab; Drug: Abemaciclib

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
Drug: Merestinib — Administered orally
  Other Names: LY2801653
  Arms: Ramucirumab + Merestinib
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Ramucirumab + Abemaciclib

SUMMARY:
The main purpose of this study is to evaluate the safety of ramucirumab in combination with other targeted agents in participants with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Study Arm 1:

  * histopathologically confirmed advanced or metastatic colorectal cancer, excluding primary tumors of appendiceal origin
  * have at least 1 measurable lesion assessable by radiological imaging. Tumor lesions located in a previously irradiated area are considered measureable if progression has been demonstrated in such lesions
  * have received prior second-line treatment with oxaliplatin and/or irinotecan, and no other licensed/standard-of-care therapies are available. If the participant has RAS wild type colorectal cancer, he or she also must have received prior treatment with an epidermal growth factor receptor monoclonal antibody
* Study Arm 2

  * pathologically confirmed mantle cell lymphoma (MCL), with (a) measurable nodal disease on positron emission tomography computed tomography (PET-CT) per Lugano classification. Prior to enrollment, pathology must be reviewed and confirmed at the investigational site where the participant is entered
  * have MCL that relapsed after or is refractory to (a) first-line combination chemotherapy with or without stem cell transplant and (b) at least 1 other locally available therapy
  * provide a newly obtained tumor tissue sample. Tumor tissue biopsies may be taken by surgical resection, core needle biopsy, or fine needle biopsy
* All Study Arms:

  * have not received previous systemic therapy (including investigational agents) targeting programmed cell death protein 1 (PD-1)/ PD-1 ligand (PDL 1) or PD-1/PDL-2 signaling pathways. Prior therapy with other immune checkpoint inhibitors, including but not limited to, anti-CD137 antibody or anticytotoxic T-lymphocyte-associated antigen-4 antibody, is not permitted
  * have adequate organ function
  * are, in the judgment of the investigator, appropriate candidates for experimental therapy after available standard therapies have failed to provide clinical benefit
  * have discontinued all previous treatments for cancer and recovered from the acute effects of therapy, other than less than or equal to Grade 2 neuropathy or nonserious and nonlife-threatening toxicities such as alopecia, altered taste, and nail changes
  * have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group scale
  * men and women must agree to the use an effective method of contraception during the study and for at least 3 months post last dose of study drug administration. Women of child-bearing potential must have negative serum and urine pregnancy tests at screening and during each treatment cycle, respectively

Exclusion Criteria:

* Study Arm 1

  * have a serious illness or medical condition including, but not limited to, the following: active or uncontrolled clinically serious infection; inadequate biliary drainage with evidence of unresolved biliary obstruction
* Study Arm 2

  * have a serious illness or medical condition including, but not limited to, the following: active or uncontrolled clinically serious infection, including chronic viral hepatitis
* All Arms:

  * have prior or concurrent malignancies, inclusive of hematologic, primary brain tumor, sarcoma, and other solid tumors, unless in complete remission with no therapy for a minimum of 5 years
  * have active gastrointestinal (GI) disease characterized by inflammatory bowel disease, malabsorption syndrome, or frequent Grade 2 or more diarrhea
  * are pregnant or breastfeeding
  * have previously documented brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression
  * have experienced any of the following: a major surgical procedure, significant traumatic injury, non-healing wound, peptic ulcer, or bone fracture less than or equal to 28 days prior to enrollment, or placement of a subcutaneous venous access device less than or equal to 7 days prior to the first dose of study treatment unless the procedure is of low risk of bleeding in the judgment of the investigator
  * have an elective or a planned major surgery during the course of the trial
  * have a known allergy or hypersensitivity reaction to any of the treatment components
  * have uncontrolled hypertension
  * have experienced any arterial thromboembolic event within 6 months prior to enrollment
  * have experienced any Grade 3 or 4 venous thromboembolic event that is considered by the investigator to be life threatening or that is symptomatic and not adequately treated by anticoagulation therapy, within 6 months prior to enrollment
  * have a history of GI perforation and/or fistulae within 6 months prior to enrollment
  * have experienced any bleeding episode considered life-threatening, or any Grade 3 or 4 GI/variceal bleeding episode in the 3 months prior to enrollment requiring transfusion or endoscopic or operative intervention
  * have congestive heart failure or poorly controlled cardiac arrhythmia per New York Heart Association Class II-IV heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs) | Cycle 1 (28 days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab, Merestinib and Abemaciclib | Predose Cycle 1 Day 1 through Predose Cycle 6 Day 1 (28 day cycles)
Proportion of Participants Who Exhibit Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)] | Baseline through Measured Progressive Disease or Death (Estimated up to 24 months)
Progression Free Survival (PFS) | Baseline through Measured Progressive Disease or Death (Estimated up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (2):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom

REFERENCES:
- [Derived] Saleh M, Cassier PA, Eberst L, Naik G, Morris VK, Pant S, Terret C, Gao L, Long A, Mao H, McNeely S, Wagner EK, Carlesi RM, Fu S. Phase I Study of Ramucirumab Plus Merestinib in Previously Treated Metastatic Colorectal Cancer: Safety, Preliminary Efficacy, and Pharmacokinetic Findings. Oncologist. 2020 Nov;25(11):e1628-e1639. doi: 10.1634/theoncologist.2020-0520. Epub 2020 Jul 17. PMID 32537847
- See also: Click here for more information about this study: A Study in Advanced Cancers Using Ramucirumab (LY3009806) and Other Targeted Agents — http://www.lillytrialguide.com/en-US/studies/advanced-cancer/JVDK#?postal=